CLINICAL TRIAL: NCT07395973
Title: The Effects of a 4-week Supplementation With a Ketogenic Nutrient Mix on 24-hour Substrate Metabolism and Muscle Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: NL-009725
Record Dates: First submitted 2025-09-08; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic nutritional supplement (Experimental): Daily ketogenic nutritional supplement for 4 weeks
  Interventions: Dietary Supplement: ketogenic nutritional Supplement
- non-ketogenic, isocaloric control (Placebo Comparator): Daily control for 4 weeks
  Interventions: Dietary Supplement: non-ketogenic, isocaloric control

INTERVENTIONS:
Dietary Supplement: ketogenic nutritional Supplement — Daily ketogenic nutritional supplement for 4 weeks
  Arms: Ketogenic nutritional supplement
Dietary Supplement: non-ketogenic, isocaloric control — Daily control for 4 weeks
  Arms: non-ketogenic, isocaloric control

SUMMARY:
This study will investigate the effect of providing a daily ketogenic nutritional supplement in the evening for a prolonged time (4 weeks) to induce a mild ketogenic state during the night in healthy elderly (60-80 years), overweight/obese (BMI: 25-35 kg/m2) individuals with low physical activity, on 24h rhythmicity in energy metabolism as compared to a non-ketogenic, isocaloric control.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60-80 years
* Body mass index (BMI) 25-35 kg/m2
* Sedentary lifestyle (not more than 2 hours of structured physical activity per week in the past 3 months)
* Stable dietary habits (no weight loss or gain > 5 kg in the past 3 months)
* Healthy (as determined by dependent physician based on medical questionnaire)
* Regular sleeping habits (7-9h of daily sleep)

Exclusion Criteria:

* Type 2 diabetes
* Participants with active congestive heart failure and/or severe renal and or liver insufficiency
* Uncontrolled hypertension
* Alcohol consumption of >3 servings per day for men and >2 servings per day for women
* Unstable body weight (weight gain or loss > 5 kg in the last 3 months) or intention to lose weight
* Participants who are on an intermittent fasting diet
* Previous enrolment in a clinical study with an investigational product during the last 3 months or as judged by the investigator which would possibly hamper our study results
* Significant food allergies/intolerance (seriously hampering study meals or study product)
* Participants who do not want to be informed about unexpected medical findings
* Blood donation during or within 2 months prior to the study
* Disturbances in circadian rhythm determined with the follow criteria:
* Extreme early bird or extreme night person (score ≤30 or ≥70 on MEQ-SA questionnaire)
* Heavily varying sleep-wake rhythm
* Night shift work during last 3 months
* Travel across > 1 time zone in the last 3 months
* High daily caffeine intake > 400mg (more than 4 cups of coffee or energy drinks)

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Delta respiratory exchange ratio (from 23:00 till 04:00) | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with indirect calorimetry

SECONDARY OUTCOMES:
Skeletal mitochondrial function | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured in muscle biopsy

OTHER OUTCOMES:
Protein and gene markers of skeletal muscle metabolism | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured in muscle biopsy
Metabolic blood markers | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured in blood samples
Interstitial ketone levels | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with a continuous ketone monitor
Interstitial glucose levels | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with a continuous glucose monitor
Whole body substrate utilization | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with indirect calorimetry
Whole body energy expenditure | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with indirect calorimetry
Physical performances | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with 6-minute walk test, chair-stand-test, and handgrip strength test
Cognitive performance | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured using Cambridge Neuropsychological Test Automated Battery (CANTAB) and cerebral perfusion measured with transcranial doppler ultrasound
Other perceivable benefits: microvasculature | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with retinal images
Other perceivable benefits: sleep quality | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with sleep quality questionnaires
Body composition | Measured after 4 weeks of daily supplementation with a ketogenic nutritional supplement or non-ketogenic, isocaloric control
  Measured with BodPod

CONTACTS AND LOCATIONS:
Overall Officials: Joris Hoeks, Dr., Principal Investigator — Maastricht University; Peter Joris, Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands